CLINICAL TRIAL: NCT05028491
Title: The Effect of Meibomian Gland Thermal Massage on Corneal Aberrations in Meibomian Gland Dysfunction Patients
Brief Title: The Influence of Meibomian Gland Expression on Corneal Aberrations in MGD Patients
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: hf-meibomian glands
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Meibomian Gland Dysfunction
Keywords: thermal massage; corneal aberrations; physical therapy
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the influence of corneal-aberrations before and after the meibomian gland thermal massage treatment.

DETAILED DESCRIPTION:
62 MGD patients treated with meibomian gland thermal massage once a week for 3 to 4 weeks were recruited.The Ocular Surface Disease Index questionnaire; tear film assessment encompassing tear meniscus height and non-invasive keratograph breakup time ; meibography score,corneal fluorescein staining; the Schirmer I test ; expressible meibomian gland, and quality ,anterior and total corneal aberrations were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* tear break-up time (BUT) ≤10 seconds or Schirmer I test (SIT) ≤10 mm, the presence of dry eye symptoms, and fluorescein staining (FL) score <3 points and at least one lid margin abnormality and poor meibomian gland expressibility

Exclusion Criteria:

* eyelid structure abnormal(Entropion , ectropion);
* having received any other treatment for MGD within three months
* history of ocular surgery
* contact lens use
* ocular infection
* any type of corneal scarring

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed as meibomian glands dysfunction in our hospital; treatment with thermal massage and expression
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
corneal aberration corneal aberrations | baseline and 1 week after treatment
  Corneal aberrations were measured with a Pentacam。 The anterior corneal wavefront aberration was expanded with normalized Zernike polynomials.The corneal aberration from 3rd to 6th order were recorded as the root mean square (RMS) for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China